CLINICAL TRIAL: NCT05670990
Title: Equine Assisted Services in Children and Adolescents With Mental Illness
Acronym: EASiCAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to methodological problems with the recruitment.
Sponsor: Peter Nymberg (Other)
Responsible Party: Sponsor-Investigator, Peter Nymberg, PhD, Halmstad University
Organization: Halmstad University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F 2022/71
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-03

CONDITIONS: Mental Disorders, Child; Mental Disorder in Adolescence; Anxiety Disorders; Anxiety; Depression; Anorexia Nervosa; School Fear
Keywords: Equine-Assisted Therapy
MeSH Terms: conditions — Neurodevelopmental Disorders; Anxiety Disorders; Depression; Anorexia Nervosa | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The randomization will take place after informed consent has been given. To achieve balance between the two groups (horse-assisted therapy or no horse-assisted therapy) we will use a minimization, so important prognostic factors are evenly distributed between the two study groups, as minimization variables we will use biological sex, age and whether the participants have contact with the child and youth psychiatry or not.
Who Masked: Investigator
Masking Description: The investigators are not involved in recruitment of the participants, and have connections to them in a roll such as employees at the recruiting locations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine assisted therapy (Experimental): once a week during 10 weeks the children will come to "Humlamaden" which is a horse farm with special trained horses and employees with specialist education in psychiatric care. During the time at the farm the child will go through a structured program that starts at the first time with just resting on the horse back under blankets
  Interventions: Other: Equine assisted therapy
- Control (No Intervention): This group will receive treatment as usual and consist of those who is randomized to control group.

INTERVENTIONS:
Other: Equine assisted therapy — A structured program that has been developed under several years at "Humlamaden" horse farm, for further information see under the description of the experimental group.
  Arms: Equine assisted therapy

SUMMARY:
Due to an increasing amount of children and adolescents are suffering from mental illnesses i Sweden. Early preventive psychological interventions are important to avoid a long-time use of medicines. Animal assisted therapy and especially equine assisted services (EAS) has shown to be a good complementary method to decrease anxiety and/or depression in children and adolescents. The main aim is to study the effect of a specific EAS program regarding symptoms of mental illness and in long-term follow-up of future healthcare consumption. We will conduct interviews with both participants and their parents besides the questionnaires at follow-ups (12 weeks, and 1 year) The intervention will be EAS at a farm following a detailed program, the staff at the farm are specially trained with a certification to practice EAS. Each session will last for about 60 minutes, once a week. Participants will get information of the study by the child and youth psychiatry in the region of Skane, and from student´s health team at elementary schools. Those who want ti participate will contact the study coordinator for full information and informed consent.

The EAS model has been used in treatment of adult with mental illness for many years, and the result are very positive. This project provides an opportunity to evaluate the effect of EAS to promote health and prevent severe manifest mental illness among children and adolescents. There are no previous studies of the long-term effect of EAS regarding health consumption.

DETAILED DESCRIPTION:
Aim and research questions The overarching aim is to evaluate the effect of EAS regarding symptoms of mental illness in both short and long-term among children and adolescents with mental illness.

The following research questions will be addressed:

Q1. What does it mean to participate in EAS for children and adolescents with mental illness and what does it mean for their parents or relatives? Q2. Does the intervention EAS lead to reduced emotional difficulties compared with control group according to children and adolescents and according to their parents or relatives? Q3. Does EAS affect conscious presence and degree of mindfulness among children and adolescents with mental illness compared with control group? Q4 Does EAS affect psychological resilience among children and adolescents with mental illness compared with control group? Q5. Are possible effects of EAS maintained up to twelve months after intervention? Q6. Are there differences in future healthcare consumption between EAS group and control group?

Study design and methods This project includes a randomized controlled trial with a longitudinal character combined with qualitative studies, to evaluate Equine Assisted Services versus no intervention.

Q1 will be answered by in-depth individual interviews with both children or adolescents and their parents or relatives.

Q2, Q3 and Q5 will captured by validated self-reported questionnaires to both children/adolescents and their parents/relatives.

Q4 and Q5 . To answer Q6, information about health care consumption will be captured from the in Health and welfare patient register, planned data outlet is planned 10 years after inclusion to study.

Participant The recruitment will be done after the child and youth psychiatry in the region of Skane in the south of Sweden, together with and the student health team at the elementary schools located nearby the horse farm, has given eligible participants notice of the study. Eligible families will be provided with oral and written information regarding the study when contacting the study coordinator. To be included the child or adolescents had to be between seven- and seventeen- years-old, with mental illness. Mental illness means in this context anxiety, depression, eating disorder, panic disorders, school refusers, and other stress related symptoms. To be included the participants must speak and understand Swedish language. The randomization will take place after informed consent has been given. To achieve balance between the two groups (horse-assisted therapy or no horse-assisted therapy) we will use a minimization, so that important prognostic factors are evenly distributed between the two study groups, as minimization variables we will use biological sex, age and whether they have contact with the child and youth psychiatry or not. The control group will receive treatment as usual.

Sample size A sample size calculation with a 1:1 relationship between two groups is estimated to a total of n=61 participants required in each group, based on a power analysis with 5% significant level and a power of 80%. Drop out is expected to be 20%. The calculation was based on other studies with horse assisted therapy [14] compared with treatment as usual, assessing depression with Spence Children's Anxiety Scale (SCAS) showing a significant difference (5.54 points) between groups. We estimate at least the same differences as in the referred study. The inclusion will be done within 3 years from the start of study.

Analysis The obtained data from interviews with the parents after 12 weeks will be analyzed by qualitative content analysis (Q1).

Interviews with children/adolescents who has participated in EAS after 12 weeks. The interviews with the children/adolescents will be based on photovoice, which gives the participants an opportunity to express what they think is important to highlight in the research. Photovoice is a method where the participants identify and choose their own starting point of the contribution to the research. The expression "Photovoice" aims to the fact that it is the participants own voice and experience which is visualised. The participants will take photographs with a digital camera during the visits at Humlamaden. The pictures should illustrate "what it implies for them to participate in EAS". The individual interviews will have starting point in the about 20 pictures with special significance for the participants. These interviews will be conducted 12 weeks after the start of EAS and twelve months after inclusion. The interviews will be recorded and start with the question "Can you tell me what the picture means to you?" During the interview, the participant narrates from without each photograph. Based on the story, clarifying and deepening questions will be asked. There will also be follow-up questions based on the analysis from previous interviews, according to Grounded Theory(Q1).

Both descriptive and analytical statistics will be used according to evaluation of any change in emotional difficulties, mindfulness, and resilience, to compare groups and for analyses of changes over time from baseline (Q2-Q6).

The intervention The twelve weeks intervention with equine assisted therapy will take place on the Humlamaden Green Rehab Foundation. The participants will visit the farm together with a parent or another relative and will be welcomed by the trained staff with an OHI-certification, issued by the organization for equine based therapy in Sweden. The trained staff will be responsible for the therapy and lead the sessions. Each session will last for about 60 minutes, once a week, and include equine based therapeutic activities. The time on the back of the horse will be conducted in a secluded and safe area, without noise or other disturbing activities, together with the certified staff . The time spent on the horse will be based on the individuals needs and conditions.The individual conditions will determine the need of eventual assistant during treatment. The horses used in therapy are specially trained for the purpose and appropriate for treatment work.

Relevance and originality The Humlamaden Green Rehab Foundation has for many years treated adults with mental illness with EAS. Together with the University of Lund and the Swedish University of Agricultural Science they have started an evaluation project of the EAS for adults at Humlamaden. Due to the patient reported positive results with EAS among adults there are many requests from parents of children with mental illness. Therefore, is it important to perform this project with focus on children and adolescents. The project will provide an opportunity to evaluate the effect of EAS to promote health and prevent severe manifest mental illness among children and adolescents. There are no previous RCTs or studies of the long-term effect (10- years) of EAS regarding health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 to 17
* Depression
* Anxiety
* School refusers
* Eating disorders
* Established contact with the child and youth psychiatry in the region of Skane
* Established contact wit the student´s health team at elementary schools in the region of Skane

Exclusion Criteria:

* Severe allergy to horses
* Do not speak, or do not understand Swedish, spoken and written.
* Do not speak, or do not understand English spoken and written.
* Those who cannot understand the intervention
* Those who do not understand what it means to be in control group

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Change in mood and feelings | 1 time each week during 14 weeks and after 12 months
  The Mood and Feelings Questionnaire, Swedish version: Short Form. 13 statements with 3 alternatives; Incorrect, Sometimes, Correct.
  Proportion of participants who change their answer between measuring points Both child and caregiver fill out the form
Mindfulness | at baseline after 14 weeks and after 12 moths
  Child Acceptance and Mindfulness Measure, Swedish version, 10 statements that shall be graded in five step scale from Never to Always.
  Proportion of participants who change their answer between measuring points
Resilience | Baseline, after 12 weeks and after 12 months
  Resilience scale, Swedish version, is a 7 graded Likert scale from Incorrect to correct, that consists of 25 statements Proportion of participants who changes their score on the scale between measuring points
Anxiety | At baseline after 14 weeks and after 12 months
  Spence Children's Anxiety Scale Swedish version, 45 statements with 4 alternatives; Never, Sometimes, Often, Always.
  Proportion of participants who change the score on the scale between measuring points
Strengths and difficulties | At baseline, after 12 weeks and after 12 months.
  Strength and Difficulties Swedish version, 25 statements with 3 alternatives; Incorrect, somewhat correct, Correct Proportion of participants who change their score on the scale between measuring points
Photovoice | 12 weeks after intervention start i.e. when the intervention ends.
  The participants will take photos by a digital camera or their own cellphone. The photos will be a starting point for a qualitative interview with each participant. Each participant will take 20 photos with a specific significant of their experience of equine assisted therapy. The following interview will be based on their photos.

SECONDARY OUTCOMES:
Compliance to intervention | during the 12 weeks of intervention
  Case report forms will be filled out regarding the participation in the intervention with equine assisted therapy Proportion of participants who follow the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nymberg, PhD, Principal Investigator — Halmstad University
Locations (1):
- Halmstad University, Halmstad, Högskolan I Halmstad, Sweden

IPD SHARING:
Plan to Share IPD: No
This is under consideration, maybe sharing after contact with PI.

REFERENCES:
- [Background] Hoagwood KE, Acri M, Morrissey M, Peth-Pierce R. Animal-Assisted Therapies for Youth with or at risk for Mental Health Problems: A Systematic Review. Appl Dev Sci. 2017;21(1):1-13. doi: 10.1080/10888691.2015.1134267. Epub 2016 Jan 25. PMID 28798541
- [Background] O'Haire ME. Animal-assisted intervention for autism spectrum disorder: a systematic literature review. J Autism Dev Disord. 2013 Jul;43(7):1606-22. doi: 10.1007/s10803-012-1707-5. PMID 23124442
- [Background] Wilson K, Buultjens M, Monfries M, Karimi L. Equine-Assisted Psychotherapy for adolescents experiencing depression and/or anxiety: A therapist's perspective. Clin Child Psychol Psychiatry. 2017 Jan;22(1):16-33. doi: 10.1177/1359104515572379. Epub 2016 Jul 27. PMID 26668260
- [Background] Schultz PN, Remick-Barlow GA, Robbins L. Equine-assisted psychotherapy: a mental health promotion/intervention modality for children who have experienced intra-family violence. Health Soc Care Community. 2007 May;15(3):265-71. doi: 10.1111/j.1365-2524.2006.00684.x. PMID 17444990
- [Background] Dimitrijevic I. Animal-assisted therapy--a new trend in the treatment of children and adults. Psychiatr Danub. 2009 Jun;21(2):236-41. PMID 19556955
- [Background] Lee PT, Dakin E, McLure M. Narrative synthesis of equine-assisted psychotherapy literature: Current knowledge and future research directions. Health Soc Care Community. 2016 May;24(3):225-46. doi: 10.1111/hsc.12201. Epub 2015 Mar 2. PMID 25727575
- [Background] Bachi K, Terkel J, Teichman M. Equine-facilitated psychotherapy for at-risk adolescents: the influence on self-image, self-control and trust. Clin Child Psychol Psychiatry. 2012 Apr;17(2):298-312. doi: 10.1177/1359104511404177. Epub 2011 Jul 14. PMID 21757481
- [Background] Beebe LH, Tian L, Morris N, Goodwin A, Allen SS, Kuldau J. Effects of exercise on mental and physical health parameters of persons with schizophrenia. Issues Ment Health Nurs. 2005 Jul;26(6):661-76. doi: 10.1080/01612840590959551. PMID 16020076
- [Background] Acil AA, Dogan S, Dogan O. The effects of physical exercises to mental state and quality of life in patients with schizophrenia. J Psychiatr Ment Health Nurs. 2008 Dec;15(10):808-15. doi: 10.1111/j.1365-2850.2008.01317.x. PMID 19012672
- [Background] Erdner A, Magnusson A. Caregivers' difficulties in activating long-term mental illness patients with low self-esteem. J Psychiatr Ment Health Nurs. 2012 Mar;19(2):140-5. doi: 10.1111/j.1365-2850.2011.01766.x. Epub 2011 Jun 22. PMID 22070619
- [Background] Berget, B., et al., Animal-Assisted Therapy with Farm Animals for Persons with Psychiatric Disorders: Effects on Anxiety and Depression, a Randomized Controlled Trial. Occupational Therapy in Mental Health, 2011. 27(1): p. 50-64.
- [Background] Holmes, C.M.P., Goodwin, D., Redhead, E.S. et al. The Benefits of Equine-Assisted Activities: An Exploratory Study. Child Adolesc Soc Work J 29, 111-122 (2012). https://doi.org/10.1007/s10560-011-0251-z
- [Background] Punzo K, Skoglund M, Carlsson IM, Jormfeldt H. Experiences of an Equine-Assisted Therapy Intervention among Children and Adolescents with Mental Illness in Sweden - A Nursing Perspective. Issues Ment Health Nurs. 2022 Dec;43(12):1080-1092. doi: 10.1080/01612840.2022.2126571. Epub 2022 Sep 30. PMID 36178465
- See also: Psychiatric care and treatment for children and young. 2019, the National Board of Health and Welfare: www.socialstyrelsen.se, December 2019. p. 118. — http://www.socialstyrelsen.se
- See also: Swedish Agency for Health Technology Assessment and Assessment of Social Services (Statens beredning för medicinsk och social utvärdering, S., Equine assisted therapy (Hästunderstödd terapi). 2019: — http://www.sbu.se/contentassets/e5a79e383f50438f8b9b73d742a623ce/hastunderstodd-terapi.pdf